CLINICAL TRIAL: NCT06100523
Title: Multidisciplinary Platform Designed to Reduce and Prevent Environmental Reprotoxic Exposures in Subfertile Couples: Assessment of the Contribution of Such Platforms on the Birth Rate After In Vitro Fertilization: Randomized Open Prospective Comparative Multicentric Study
Brief Title: PREVenting-ENvIronment-Reprotoxic Exposures Before In Vitro Fertilization (PREVENIR-FIV)
Acronym: PREVENIR-FIV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RCAPHM21_0387; 2022-A01017-36 (Other: ID RCB)
Record Dates: First submitted 2023-09-21; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-09

CONDITIONS: Infertility
Keywords: Infertility; In Vitro Fertilization; Intracytoplasmic Sperm Injection
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (interventional) (Experimental): Analysis of the responses to the self-administered questionnaires with, if necessary, protocol interview concerning environmental and occupational factors, which will determine the consultations to be planned for their follow-up by the platform
  Interventions: Behavioral: Visioconsulation; Biological: hair sampling; Behavioral: self-assessment questionnaire on dedicated application; Behavioral: Specialized follow-up; Behavioral: self-assessment questionnaire for follow-up
- Arm B (standard management) (Active Comparator): Care path according to the usual modalities of the assisted reproductive treatment (ART) center
  Interventions: Behavioral: self-assessment questionnaire; Biological: hair sampling; Behavioral: self-assessment questionnaire for follow-up

INTERVENTIONS:
Behavioral: Visioconsulation — Meeting by videoconsultation with professionals adapted to the exposures highlighted by the questionnaires for patients who responded on the dedicated application (Arm A)
  Arms: Arm A (interventional)
Behavioral: self-assessment questionnaire — self-administered questionnaire of assessment of reprotoxic exposures, assessment of stress, physical activity, quality of life in infertility course
  Arms: Arm B (standard management)
Biological: hair sampling — hair sampling from the 2 members of the couple
Behavioral: self-assessment questionnaire on dedicated application — self-administered questionnaire of assessment of reprotoxic exposures, assessment of stress, physical activity, quality of life in infertility course
  Arms: Arm A (interventional)
Behavioral: Specialized follow-up — proactive healthcare pathway : active support of corrective measures implemented with couples by the platform, with the help of the application
  Arms: Arm A (interventional)
Behavioral: self-assessment questionnaire for follow-up — self-administered questionnaire of assessment of reprotoxic exposures, assessment of stress, physical activity, quality of life in infertility course

SUMMARY:
The objective is to evaluate the effectiveness of an innovative personalized management strategy adapted to the level of environmental risk, in a population of infertile couples, eligible for assisted reproductive treatment (ART) by intraconjugal In Vitro Fertilization (IVF)/ Intracytoplasmic sperm injection (ICSI).

Consultation of the couple at the ARTcenter : - Prescriptions of the standard assessment of infertility to the couples eligible for ART. - Inclusion and randomization (arm A interventional vs arm B standard management) of the couples having signed the consent. - Information for each patient on a standardized online self questionnaire on environmental exposures, physical activity and stress.

DETAILED DESCRIPTION:
* Arm A (interventional): analysis of the responses to the self-administered questionnaires with, if necessary, protocol interview concerning environmental and occupational factors, which will determine the consultations to be planned for their follow-up by the platform. - support of couples by the multidisciplinary platform with the help of the downloaded application: Meeting by videoconsultation with professionals adapted to the exposures highlighted by the questionnaires. Multidisciplinary Synthesis (MS): Synthesis of the first consultations and the results of the self-questionnaires by the multidisciplinary team. Determination of preventive and corrective measures, specific advice, specialized follow-up if necessary. Presentation to patients of the personalized measures decided in MS: information on the personalized management proposed (follow-up addictologist, dietician, psychologist, occupational doctor), personalized advice sheets. Couples who do not require personalized measures will continue their treatment with prevention advice adapted to their profession and their environment. Transmission of the minutes of the MS to the clinician in charge of the couple.
* Arm B (standard management): care path according to the usual modalities of the ART center (indications, network of practitioners, monitoring and information tools). If necessary, distribution by the clinician of information leaflets on addictions, dietetics + distribution of a general information leaflet on reprotoxic factors.

In both arms: embryology consultation before ART: information on the planned ART. Information on the online self-assessment questionnaire for assessing reprotoxic exposures, assessing stress, physical activity, and quality of life during infertility. In centers with a biological resource center Germethèque, hair sampling from the 2 members of the couple.

First attempt of IVF/ICSI, in both arms, followed for 24 months with every 6 months: information of the online self-administered questionnaire of assessment of reprotoxic exposures, assessment of stress, physical activity, quality of life in infertility course. At 12 months and 24 months: hair sampling from both members of the couple (in Germethèque centers only).

- In arm A during the 24 months of follow-up: active support of corrective measures implemented with couples by the platform, with the help of the application (weight loss goals, changes in habits, physical activity, decreased or stopped toxics). Continuation of specialized follow-up if necessary, in videoconsultation.

At the end of the study: a sample of about twenty couples in each arm will be the subject of a semi-directed interview aimed at qualitatively determining the brakes and levers to their adherence to the environmental health advice received during their management in ART.

Medical-economic analysis: a cost-effectiveness analysis and a budget impact analysis will be carried out by the Epidemiology and Health Economics Department.

ELIGIBILITY:
Inclusion Criteria:

* Couple eligible for a first attempt of conventional In Vitro Fertilization (IVF) or Intra Cytoplasmic Sperm Injection (IVF-ICSI) intra-marital;
* Signature of informed consent by both partners of the couple;
* Possession of a smartphone.

Exclusion Criteria:

* Not fluent in the language;
* Refusal to participate in the study of one or both members of the couple;
* Use of cryopreserved intra-conjugal gametes before management in MPA;
* Use of gamete donation, embryo reception;
* History of chemotherapy/radiotherapy;
* Support in viral risk circuit;
* Not having a smartphone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4224 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Clinical live birth rate | 24 months
  Proportion of couples who obtained at least one live birth during the 24 months of assisted reproductive treatment (ART) treatment (birth(s) obtained after In Vitro Fertilization (IVF)/Intracytoplasmic Sperm Injectionc (ICSI), frozen embryo transfer (FET) from IVF/ICSI, or spontaneous pregnancy obtained between ART treatments), in Arm A versus arm B.

SECONDARY OUTCOMES:
Clinical pregnancy rate | 24 months
  Proportion of couples who achieved at least one clinical pregnancy (presence of gestational sac with cardiac activity at 8 SA) during the 24 months of ART management (pregnancies obtained after IVF/ICSI, frozen embryo transfers (FET) or spontaneously), comparison in both arms.
Embryology markers | 24 months
  In IVF/ICSI performed in both arms, comparison of fertilization rates, rate of useful embryos (transferred or cryopreserved), embryo implantation rate
Pregnancy markers | 24 months
  On clinical pregnancies obtained after ART or spontaneously during the 24 months of ART management, comparison in both arms: rates of progressive pregnancies (presence of cardiac activity at 12 weeks of amenorrheae)
Pregnancy markers | 24 months
  On clinical pregnancies obtained after ART or spontaneously during the 24 months of ART management, comparison in both arms: rates of obstetric pathology (at least one of the following complications = high blood pressure, gestational diabetes, cholestasis, placenta previa, placental abruption, intrauterine growth retardation, missing twin syndrome, premature rupture of membranes, threat of premature delivery, 3rd trimester hemorrhage, preterm birth, postpartum hemorrhage)
Newborn health | at birth
  term,
Behavior changes | 24 months
  evaluation of behavior changes like : consumption of toxic substances, physical activity, eating habits, stress management, protection against environmental/occupational reprotoxins and the quality of life of couples in both arms during follow-up
qualitative analysis | 24 months
  Qualitative analysis of the brakes and levers related to the adherence of couples to the measures of prevention and correction of reprotoxic exposures proposed during their management in ART (in both arms)

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Director — Assistance Publique - Hôpitaux de Marseille
Locations (1):
- Assitance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sunyach C, Courbiere B, Simon N, Delva F, Garlantezec R, Bretelle F, Leandri R, Gehanno JF, Esquirol Y, Loubiere S, Resseguier N, Sari-Minodier I, Perrin J. PREVENIR-IVF: study protocol for a prospective multicentre randomized open comparative trial, which explores the efficacy of a multidisciplinary platform reducing and preventing reprotoxic environmental exposures in subfertile couples on live birth rate after assisted reproduction treatment. Trials. 2025 Dec 22;26(1):575. doi: 10.1186/s13063-025-09208-8. PMID 41430276